CLINICAL TRIAL: NCT03795727
Title: Clinical Evaluation of Sectional Matrix Versus Circumferential Matrix for Reproduction of Proximal Contact by Undergraduate Students and Postgraduate Dentists: Randomized Controlled Trial
Brief Title: Clinical Evaluation of Sectional Matrix Versus Circumferential Matrix for Reproduction of Proximal Contact
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Omar Osama Shaalan, Lecturer of conservative dentistry, Faculty of Dentistry, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: circumferential vs sectional
Record Dates: First submitted 2019-01-03; First posted 2019-01-08 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Proximal Contact

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sectional matrix (Experimental): precontoured sectional matrix band
  Interventions: Device: MD ring and precontoured sectional matrix by TOR VM
- Circumferential matrix (Active Comparator): Circumferential matrix band applied by tofflemire retainer
  Interventions: Device: Circumferential matrix and tofflemire retainer by Kerr

INTERVENTIONS:
Device: MD ring and precontoured sectional matrix by TOR VM — MD ring (separation ring) and precontoured sectional matrix (thickness 0.035mm hard) and a wedge was used to secure matrix in place
  Arms: Sectional matrix
Device: Circumferential matrix and tofflemire retainer by Kerr — Circumferential matrix (thickness 0.038mm) applied by tofflemire retainer and secured in place with wedge
  Arms: Circumferential matrix

SUMMARY:
The aim of this study is to evaluate the effects of different matricing techniques either sectional matrix or circumferential matrix on reproduction of optimum proximal contacts and contours during restoration of class II cavities with resin composite by undergraduate students or postgraduate dentists.

ELIGIBILITY:
Inclusion Criteria:

* Compound class II cavities
* Good oral hygiene
* No spacing or crowding
* Healthy peridontium

Exclusion Criteria:

* Complex class II cavities
* Poor oral hygiene
* Spacing or crowding
* Evidence of peridontal disease

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2020-01-20 (Actual); Primary Completion 2020-02-12 (Actual); Study Completion 2020-03-12 (Actual)

PRIMARY OUTCOMES:
Proximal contact | Up to 3 hours from randomization till contact is restored
  Reproduction of proximal contact either optimum, tight or loose (Categorical)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Cairo University, Cairo, El Manial, Egypt

IPD SHARING:
Plan to Share IPD: No